CLINICAL TRIAL: NCT02138266
Title: Comparative Study of the Topcon Specular Microscope SP-1P and the Konan Specular Microscope CELLCHEK XL (Predicate Device) for the Measurements of Endothelial Cell Density Measurements, Coefficient of Variation of Endothelial Cell Area, ％ Hexagonality, Central Corneal Thickness
Brief Title: Comparative Study of Specular Microscopes for Endothelial and Corneal Cell Measurements
Status: Completed | Type: Observational
Sponsor: Topcon Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Organization: Topcon Corporation (Industry)
Other Study IDs: TOPCON-SP-1P-US-0001
Record Dates: First submitted 2014-05-05; First posted 2014-05-14 (Estimated); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Corneal Endothelial Cell Loss
MeSH Terms: conditions — Corneal Endothelial Cell Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Non-Pathologic Adults age 18-28 yrs: Non-Pathologic Adults age 18-28 yrs
  Interventions: Device: Topcon Specular Microscope SP-1P; Device: Konan Specular Microscope CELLCHEK XL
- Non-Pathologic Adults age 29-80 yrs: Non-Pathologic Adults age 29-80 yrs
  Interventions: Device: Topcon Specular Microscope SP-1P; Device: Konan Specular Microscope CELLCHEK XL
- Pathologic Adults age 29-80 yrs: Pathologic Adults age 29-80 yrs
  Interventions: Device: Topcon Specular Microscope SP-1P; Device: Konan Specular Microscope CELLCHEK XL

INTERVENTIONS:
Device: Topcon Specular Microscope SP-1P
Device: Konan Specular Microscope CELLCHEK XL

SUMMARY:
The primary objective of this clinical study is to collect clinical data to support an FDA 510(k) submission for the Topcon Specular Microscope SP-1P. The secondary objective is to evaluate any adverse events found during the clinical study.

ELIGIBILITY:
Inclusion Criteria -Non-Pathologic Young Adults (18-28 years old) and Non-Pathologic Adults (29-80 years old):

* Male or female subjects from 18 to 80 years old who have full legal capacity to volunteer on the date the informed consent is signed;
* Subjects who can follow the instructions by the clinical staff at the clinical site, and can attend examinations on the scheduled examination date;
* Subjects who agree to participate in the study.

Inclusion Criteria -Pathologic Adults (29-80 years old)

* Male and female subjects from 29 to 80 years old who have full legal capacity to volunteer on the date the informed consent is signed;
* Subjects who can follow the instructions by the clinical staff at the clinical site, and can attend examinations on the scheduled examination date;
* Subjects who agree to participate in the study;
* At least one eye with any of the following conditions:

  * History of post-op surgical trauma including Pseudophakic or Aphakic bullous keratopathy;
  * History of corneal transplant;
  * Physical injury or trauma to the cornea;
  * Long term Fuch's dystrophy/Guttata (and other corneal endothelial dystrophies)
  * Keratoconus;
  * Long term PMMA contact lens use (greater than 3 years).

Exclusion Criteria -Non-Pathologic Young Adults (18-28 years old) and Non Pathologic Adults (29-80 years old)

* History of corneal transplant;
* Long term Fuch's dystrophy (and other corneal endothelial dystrophies);
* Keratoconus;
* Guttata;
* Diabetes mellitus type I or type II;
* History of cataract, refractive or ocular surgical procedures that render the cornea opaque or otherwise impact its ability to be imaged using the investigational device;
* All contact lens wearers;
* Fixation problems which may prevent obtaining good quality SP-1P and CELLCHEK PLUS in either eye.

Exclusion Criteria -Pathologic Adults (29-80 years old):

* Fixation problems which may prevent obtaining at least poor quality (refer to Figure 1) SP-1P and KONAN CELLCHEK PLUS images in either eye.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ophthalmology Practice
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2014-02; Primary Completion 2014-03 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Corneal endothelial cell density | Single time point - 1 day
Coefficient of variation of endothelial cell area | Single time point - 1 day
Corneal endothelial cell % hexagonality | Single time point - 1 day
Central corneal thickness | Single time point - 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States